CLINICAL TRIAL: NCT02546583
Title: Diagnosing and Targeting Mechanisms of Diuretic Resistance in Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1505015805; 1R01HL128973-01 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-09-11 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Bumetanide; Furosemide; Chlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Increased Intravenous Loop Diuretic (Bumetanide or Furosemide) (Experimental): 2.5x Visit 1 dose
  Interventions: Drug: Increased Intravenous Bolus Loop Diuretic Dose (Bumetanide or Furosemide)
- Loop Diuretic (Bumetanide or Furosemide) + IV Chlorothiazide (Experimental): Loop diuretic (Bumetanide or Furosemide) dose remains the same as visit 1 dose but now with the addition of 500-1000 mg IV chlorothiazide
  Interventions: Drug: IV Chlorothiazide
- Observational Arm (No Intervention): Subjects taking an IV loop diuretic (Bumetanide or Furosemide) that have sodium output greater than 100 mmol. These subjects will continue to be followed and have data collected on them.

INTERVENTIONS:
Drug: Increased Intravenous Bolus Loop Diuretic Dose (Bumetanide or Furosemide) — An increase to 2.5x the Visit 1 dose of loop diuretic (bumetanide or furosemide).
  Arms: Increased Intravenous Loop Diuretic (Bumetanide or Furosemide)
Drug: IV Chlorothiazide
  Arms: Loop Diuretic (Bumetanide or Furosemide) + IV Chlorothiazide

SUMMARY:
Effective diuresis is the primary goal of most acute decompensated heart failure hospitalizations, but diuretic resistance is common and our ability to detect it is limited. Further, there are therapeutically distinct groups of diuretic-resistant patients. These are not easily distinguished using currently available methods, leading to trial-and-error based treatment that promotes lengthy hospitalizations.

The aims of this study are:

1. To develop inexpensive and efficient tools to predict diuretic response
2. To understand the prevalence of therapeutically targetable mechanisms of diuretic resistance using endogenous lithium clearance
3. To develop methodology to differentiate diuretic resistance mechanisms using common/inexpensive laboratory tests
4. To provide proof of concept that mechanistically tailored diuretic therapy can improve natriuresis

DETAILED DESCRIPTION:
This study is a minimal-risk observational open-label single center study with randomization between two standard of care interventions. Approximately 500 patients admitted to the hospital (Yale New Haven Health System) with a clinical diagnosis of heart failure will be enrolled in the overall study.

Patients will undergo sampling of their blood and collection of urine at a minimum of 4 timepoints (called "visits"), or a minimum of 5 in the interventional arm. Patients with a low urine sodium output (<100 mmol) on Visit 1 will be eligible for 1:1 randomization to either an increased dose of their Visit 1 loop diuretic or addition of IV chlorothiazide to their Visit 1 loop diuretic.

ELIGIBILITY:
For all patients:

Inclusion criteria:

* Age ≥ 18 years
* Clinical diagnosis of ADHF with at least one objective sign of volume overload: rales, edema, elevated JVP, preadmission weight gain
* Current use of bolus IV loop diuretic therapy and projected need by the treating clinician for continued treatment with IV diuretics for at least 3 days with the goal of significant fluid removal (>1L net fluid loss/day)

Exclusion criteria:

* Inability to perform informed consent or comply with the serial urine collection procedures
* Significant bladder dysfunction or urinary incontinence
* Hematocrit less than 21% or active bleeding

For patients in the interventional arm:

Inclusion criteria:

* Cumulative 6-hour sodium output < 100 mmol following Visit 1 IV loop diuretic dose
* Visit 1 IV loop diuretic dose ≤ 160 mg of furosemide equivalents
* Serum sodium > 125 mmol/L
* At least 6 hours since last dose of diuretic

Exclusion criteria:

* Current use or projected future requirement by the treating physician for thiazide diuretics
* Use of high dose mineralocorticoid receptor antagonist therapy (>50mg of spironolactone or >100mg of eplerenone) or amiloride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Accuracy of sodium prediction equation in predicting suboptimal natriuretic response to a dose of diuretics | 6 hours
  Suboptimal Natriuretic Response is defined as a measured sodium output of <100 mmol in the 6 hours following the dose of diuretic
Prevalence of mechanistic sub types of Diuretic Resistance (DR) as defined by cutoff values of change in fractional excretion of lithium | 6 hours
  Descriptions of the prevalence of the DR mechanisms at the different time points in the study will be reported.
Accuracy of prediction of mechanistic sub types of DR using universally available laboratory tests | 6 hours
  The relationship between the change in fractional excretion of potassium and sodium and the change in fractional excretion of endogenous lithium will be assessed in order to develop methodology to identify the etiology of DR using universally available laboratory tests.
Change in total 6-hour sodium output between observational and randomized intervention study days, compared between intervention groups | 6 hours
  Sodium output in response to a dose of diuretics will be measured via urine collection.

SECONDARY OUTCOMES:
Prediction of mechanistic sub types of DR | 6 hours
  Relationship between the fractional excretion of magnesium or calcium with the fractional excretion of endogenous lithium will also be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Rao VS, Cox ZL, Ivey-Miranda JB, Moreno-Villagomez J, Ramos-Mastache D, Maulion C, Bellumkonda L, Turner J, Wilson FP, Shilpak MG, Estrella MM, Welling P, Wilcox CS, Ellison DH, Forbush B, Testani JM. Loop Diuretic Dose Intensification versus Adjuvant Thiazide for Diuretic Resistance in Acute Heart Failure: Mechanistic Randomized Controlled Trial. J Am Soc Nephrol. 2025 Sep 12. doi: 10.1681/ASN.0000000887. Online ahead of print. No abstract available. PMID 40938670
- [Derived] Ivey-Miranda JB, Rao VS, Cox ZL, Moreno-Villagomez J, Mahoney D, Maulion C, Bellumkonda L, Turner JM, Collins S, Wilson FP, Krumholz HM, Testani JM. In-Hospital Observation on Oral Diuretics After Treatment for Acute Decompensated Heart Failure: Evaluating the Utility. Circ Heart Fail. 2023 Apr;16(4):e010206. doi: 10.1161/CIRCHEARTFAILURE.122.010206. Epub 2023 Mar 10. PMID 36896716